CLINICAL TRIAL: NCT02988492
Title: Acute Stroke Thrombectomy: Does CT Perfusion Accurately Predict Infarct on MRI After Recanalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MR-RETRIEVE Protocol
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI perfusion imaging (Other): MRI screening will be performed as per standard-of-care by the MRI technologist staff. Imaging will be performed with 1.5 T or 3 T systems (Magnetom Vision; Siemens, Erlangen, Germany) using a multisection, single shot, spin echo, echo planer imaging sequence. Diffusion gradients will be applied in each of the x, y and z directions with three b values (0, 500 and 1000 s/mm2). Imaging parameters include a TE of 94 ms, field of view of 23 cm, matrix of 128 and section thickness of 5.5 mm for the 1.5 T system and a TE of 83 ms, field of view of 23 cm, matrix of 128 and section thickness of 3 mm for the 3 T system. Conventional spin echo imaging also will be performed at each examination under T1 and T2 weighted conditions, with a fluid attenuated inversion recovery sequence and Time-of-flight MRA of the Circle-of-Willis.
  Interventions: Device: MRI perfusion imaging

INTERVENTIONS:
Device: MRI perfusion imaging — Evaluate the sensitivity and specificity of whole---brain CTP in predicting 24 hour DWI---MRI infarct in patients with acute proximal anterior circulation occlusions successfully recanalized with endovascular treatment.

SUMMARY:
The newest generation of stent---retrievers results in higher recanalization rates and faster recanalization time compared to older generation endovascular therapies for acute stroke. Advanced neuroimaging can potentially improve the assessment of infarct core and inform decision---making in patients being considered for endovascular therapy. Evaluation of infarct core may be performed with NECT, CTASI or CT perfusion. In the past, evaluation of CTP in predicting core infarct in acute stroke has been limited because recanalization status was lacking. In addition, final infarct size may be underestimated on NECT compared with MRI. These two limitations can now be addressed: the new generation of stent---retrievers allows accurate determination recanalization time; evaluating the test characteristics of CTP using 24 hour DWI---MRI as the reference standard can be readily performed.

We aim to prospectively investigate the sensitivity and specificity of whole---brain CTP in predicting 24 hour DWI---MRI infarct in patients with acute proximal anterior circulation occlusions successfully recanalized with endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Admission NECT, CTA neck and COW or multi-phase CTA or CTP. Follow---up 24 hr DWI---MRI performed
2. Endovascular therapy performed for acute anterior circulation stroke as per clinical practice.
3. Patient with an angiographically documented ICA, M1 or M2 occlusion

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the sensitivity and specificity of CTP | Up to 24 months
  The primary outcome of our study is to evaluate the sensitivity and specificity of CTP in predicting infarct on 24 hour DWI---MRI.

SECONDARY OUTCOMES:
Correlate advanced imaging to clinical outcome | Up to 24 months
  The secondary outcome of our study is to correlate advanced imaging to clinical outcome at 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Iancu, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided